CLINICAL TRIAL: NCT00260065
Title: A Phase 2 Study of Decitabine Administered Daily for 5 Days Every 4 Weeks to Adults With Advanced-Stage Myelodysplastic Syndromes
Brief Title: A Study of Decitabine Given to Adults With Advanced-Stage Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACO-020
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2010-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Decitabine; Dacogen; MGI Pharma
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20mg/m^2, IV on days 1-5 of each 28 day cycle; until progression, death or unacceptable toxicity develops.
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to determine the overall response rate in patients with myelodysplastic syndromes (MDS) given a daily dosing schedule of decitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an Institutional Review Board (IRB) -approved informed consent form.
2. Must be 18 years of age or older.
3. Must have a diagnosis for MDS fitting any of the recognized French-American-British (FAB) classifications and International Prognostic Scoring System (IPSS) greater than or equal to 0.5 as determined by Complete Blood Count (CBC), bone marrow assessment, and cytogenetics within 28 days of receiving study drug. If FAB classification is Refractory anemia (RA) or Refractory anemia with ringed sideroblasts (RARS), then must be red cell transfusion dependent, defined as needing red cells more frequently than once every 4 weeks.
4. If receiving erythropoietin(Procrit), must have been on a stable dose for at least 8 weeks before first dose of study drug.
5. If receiving darbepoetin(Aranesp), must have been on a stable dose for at least 12 weeks before first dose of study drug.

Exclusion Criteria:

1. Must not have a diagnosis of Acute Myeloid Leukemia (AML) or other progressive malignant disease.
2. Must not have received any investigational agent within the 30 days preceding the first dose of study drug.
3. Must not have uncontrolled cardiac disease or uncontrolled congestive heart failure.
4. Must not have an active viral or bacterial infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Inc.
Locations (21):
- United States (20):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Boca Raton, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Griffin, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Rochester, Minnesota
  - Hackensack, New Jersey
  - Buffalo, New York
  - Canton, Ohio
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Houston, Texas
  - Midland, Texas
  - Seattle, Washington
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
- Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jabbour E, Kantarjian H, O'Brien S, Kadia T, Malik A, Welch MA, Teng A, Cortes J, Ravandi F, Garcia-Manero G. Retrospective analysis of prognostic factors associated with response and overall survival by baseline marrow blast percentage in patients with myelodysplastic syndromes treated with decitabine. Clin Lymphoma Myeloma Leuk. 2013 Oct;13(5):592-6. doi: 10.1016/j.clml.2013.05.004. Epub 2013 Jun 20. PMID 23790798
- [Derived] Jabbour E, Garcia-Manero G, Ravandi F, Faderl S, O'Brien S, Fullmer A, Cortes JE, Wierda W, Kantarjian H. Prognostic factors associated with disease progression and overall survival in patients with myelodysplastic syndromes treated with decitabine. Clin Lymphoma Myeloma Leuk. 2013 Apr;13(2):131-8. doi: 10.1016/j.clml.2012.11.001. Epub 2012 Dec 21. PMID 23260600
- See also: MGI Pharma's website — http://www.mgipharma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine 20 mg/m2 Intravenous: Decitabine 20 mg/m2 intravenous IV on Days 1-5 of each 28 day cycle.
Period: Overall Study
Arm/Group | Decitabine 20 mg/m2 Intravenous
Started | 99
Completed | 6
Not Completed | 93
Not completed — Progressive Disease | 22
Not completed — Adverse Event | 17
Not completed — Death | 13
Not completed — Withdrawal by Subject | 13
Not completed — Physician Decision | 19
Not completed — Not otherwise specified | 8
Not completed — Medication Noncompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine 20 mg/m2 Intravenous
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 70.9 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 86
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Overall Response
Description: Overall Response = complete remission (disappearance of all target lesions) + partial remission (at least 30% decrease in the sum of the longest diameters of target lesions)
Time Frame: 1 year
Population: Intent-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Decitabine 20 mg/m2 Intravenous
Number analyzed (Participants) | 99
participants | 33
Statistical Analysis 1: Comparison: Decitabine 20 mg/m2 Intravenous; Test type: Superiority or Other; Percentage of Participants = 33, 95% CI [24.2 to 43.5]

2. Secondary Outcome: Best Response and Overall Improvement
Description: Overall Improvement = complete remission + marrow complete remission + partial remission + hematologic improvement (CR+mCR+PR+HI)
Time Frame: 1 year
Population: Intent-to-treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Decitabine 20 mg/m2 Intravenous
Number analyzed (Participants) | 99
Participants
  Overall Improvement | 51
  Complete Remission (CR) | 17
  Marrow Complete Remission (mCR) | 16
  Partial Remission (PR) | 0
  Hematologic Improvement (HI) | 18
Statistical Analysis 1: Comparison: Decitabine 20 mg/m2 Intravenous; Test type: Superiority or Other; Percentage of Participants = 52, 95% CI [41.3 to 61.7]

ADVERSE EVENTS:
Arm/Group | Decitabine 20 mg/m2 Intravenous
Serious Adverse Events (participants affected / at risk) | 65/99
Other Adverse Events (participants affected / at risk) | 96/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m2 Intravenous (N=99)
Anaemia (Blood and lymphatic system disorders) | 9
Febrile Neutropenia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 12
Pancytopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiac Failure Congestive (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Disease Progression (General disorders) | 4
Pyrexia (General disorders) | 6
Cellulitis (Infections and infestations) | 2
Clostridial Infection (Infections and infestations) | 3
Lung Infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 17
Sepsis (Infections and infestations) | 4
Septic Shock (Infections and infestations) | 2
Staphylococcal Bacteraemia (Infections and infestations) | 7
Staphylococcal Sepsis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m2 Intravenous (N=99)
Anaemia (Blood and lymphatic system disorders) | 31
Febrile Neutropenia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 38
Pancytopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 27
Thrombocythaemia (Blood and lymphatic system disorders) | 5
Cardiac Failure Congestive (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 8
Ear Pain (Ear and labyrinth disorders) | 6
Abdominal Pain (Gastrointestinal disorders) | 14
Abdominal Pain Upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 30
Diarrhea (Gastrointestinal disorders) | 28
Dyspepsia (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 5
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 40
Oral Pain (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 11
Toothache (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 15
Chest Pain (General disorders) | 6
Chills (General disorders) | 16
Fatigue (General disorders) | 46
Mucosal Inflammation (General disorders) | 9
Oedema (General disorders) | 5
Oedema Peripheral (General disorders) | 27
Pain (General disorders) | 5
Pyrexia (General disorders) | 36
Cellulitis (Infections and infestations) | 9
Oral Candidiasis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 20
Sinusitis (Infections and infestations) | 6
Staphylococcal Bacteraemia (Infections and infestations) | 8
Tooth Abscess (Infections and infestations) | 5
Upper Respiratory Tract Infection (Infections and infestations) | 10
Urinary Tract Infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 9
Blood Bilirubin Increased (Investigations) | 6
Breath Sounds Abnormal (Investigations) | 5
Weight Decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 23
Decreased Appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 18
Bone Pain (Musculoskeletal and connective tissue disorders) | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 18
Anxiety (Psychiatric disorders) | 9
Confusional State (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 5
Night Sweats (Skin and subcutaneous tissue disorders) | 5
Petechiae (Skin and subcutaneous tissue disorders) | 12
Pruritis (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 11
Skin Lesion (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 11
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No